CLINICAL TRIAL: NCT00041431
Title: Estrogen, Cytokines and Heart Failure in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double
Other Study IDs: 1181; R01HL068939 (NIH)
Record Dates: First submitted 2002-07-08; First posted 2002-07-09 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2005-05

CONDITIONS: Cardiovascular Diseases; Heart Failure, Congestive; Heart Diseases; Menopause
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure; Heart Diseases | interventions — Hormone Replacement Therapy

INTERVENTIONS:
Drug: Hormone Replacement Therapy

SUMMARY:
To determine the effects of estrogen therapy on postmenopausal women with congestive heart failure.

DETAILED DESCRIPTION:
BACKGROUND:

Congestive heart failure (CHF) is a leading cause of morbidity, mortality, and hospitalization in women. The increase in mortality suggests that postmenopausal estrogen loss may alter the phenotypic expression of CHF. Because estrogen is a potent in vitro inhibitor of pro-inflammatory cytokines (e.g., TNFa, IL-1B, IL-6), which are re-expressed by the failing myocardium in patients with CHF and are related to an adverse prognosis, the study postulates that estrogen replacement will improve the outcome of postmenopausal women with CHF.

DESIGN NARRATIVE:

The randomized, double blind study was conducted in 166 postmenopausal women with congestive heart failure due to idiopathic (i.e.nonischemic) dilated cardiomyopathy and NYHA class II or III symptoms on either combined estrogen and progestin or placebo. Women maintained their then current congestive heart failure medications for six months. Three outcomes were measured: 1) Congestive heart failure severity/functional capacity quantified by maximum oxygen consumption during metabolic stress testing; 2) Left and right ventricular remodeling quantified by electron bean CT scan; 3) quality of life assessment by the Minnesota Living with Heart Failure and Kansas City cardiomyopathy questionnaires. In addition, measurements were made of pro-inflammatory markers, that had been demonstrated to be elevated in congestive heart failure to assess whether hormone replacement therapy reduced them.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Postmenopausal women with NYHA Class II or Class III congestive heart failure due to idiopathic dilated cardiomyopathy.

Max Age: 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-12; Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Reis — University of Pittsburgh